CLINICAL TRIAL: NCT02824588
Title: Executive Control, Processing Speed and Memory Function in Long- Term Peripheral Neuropathic Pain and Fibromyalgia
Brief Title: Working Memory Training for Chronic Neuropathic and Fibromyalgia Pain
Acronym: NEPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Henrik Børsting Jacobsen, Post Doctoral Fellow, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016/8442
Record Dates: First submitted 2016-06-27; First posted 2016-07-06 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Working Memory Deficits; Neuropathic Pain; Fibromyalgia
Keywords: Pain; Working memory
MeSH Terms: conditions — Neuralgia; Fibromyalgia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Working Memory Training
  Interventions: Behavioral: Working Memory Training
- Control (Active Comparator): Internet use
  Interventions: Behavioral: Internet use

INTERVENTIONS:
Behavioral: Working Memory Training — Training mental flexibility
  Arms: Intervention
Behavioral: Internet use — Used as control for time spent on computer
  Arms: Control

SUMMARY:
The goal of this project is to investigate and improve executive control function in two distinct pain conditions, namely neuropathic pain and fibromyalgia (FM). It is hypothesized that there is a significant difference in the executive control function of patients with neuropathic pain and FM pain. It is also hypothesized that all participants with poor executive control functioning will report significant improvements in pain intensity, functioning and cognitive complaints following cognitive training. The study tests and influence the working memory concepts of inhibition, updating and flexibility through an experimental, cross-over treatment design.

To perform the experiment, we will recruit 160 participants (80 with neuropathic pain and 80 with FM) from the Departments of pain management and research at St Olav's University Hospital and Oslo University Hospital (OUS). The proposed design will be able to determine whether or not executive control, processing speed and memory function differs in two distinct populations of pain patients. Moreover, whether impairments are amended by computerized training.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of fibromyalgia or neuropathic pain
* Confirmed objective cognitive impairments on the CANTAB battery compared to IQ control

Exclusion Criteria:

* Mania, suicidal ideation and/or active psychosis
* No objective cognitive impairments
* Personality disorders
* Pregnancy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Objective neuropsychological tests | 36 weeks
  CANTAB test battery

SECONDARY OUTCOMES:
Pain intensity | 36 weeks
  VAS scale
Stress regulation | 36 weeks
  Hair cortisol
Symptoms of depression | 36 weeks
  Hopkins symptom checklist
Sleep duration, quality and awakening | 36 weeks
  Actigraphy
Quality of life | 36 weeks
  EQ-5D
Medication use | 36 weeks
  Registered analgetic usage
Self-reported memory and concentration impairments | 36 weeks
  Everyday Memory Questionnaire
Self-reported cognitive intrusion | 36 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway